CLINICAL TRIAL: NCT03385291
Title: Effects of Acoustic Stimuli in Patients With Disorders of Consciousness: An Electroencephalography and Neuroimaging Study
Brief Title: Effects of Different Stimuli in Patients With Disorders of Consciousness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: disorders of consciousness
Record Dates: First submitted 2017-10-24; First posted 2017-12-28 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2017-10

CONDITIONS: Disorder of Consciousness
Keywords: EEG;DOC;auditory
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with disorders of consciousness (Experimental): 3 minutes stimulation with music,name,and noise separately,each are separated with a 5 minutes washout period.
  Interventions: Device: music,name,and noise sound
- healthy control group (Experimental): 3 minutes stimulation with music,name,and noise separately,each are separated with a 5 minutes washout period.
  Interventions: Device: music,name,and noise sound

INTERVENTIONS:
Device: music,name,and noise sound — A 5-minute baseline silence was followed by the presentation of three contrasting auditory stimuli(music,name,and noise), with a 2-minute washout silence separating each stimulus

SUMMARY:
In recent years, promoting wakening attempts in patients with disorders of consciousness are increasing, but there are a lack of objective indicators to evaluate the efficacy and further researches on the brain mechanism during the wakening processing. So, the study first assessed the cerebral response during emotional acoustic stimuli with quantitative EEG and ERP(Event-related potential), and next, the investigators explored the relationship between brain activation and patients' recovery.

DETAILED DESCRIPTION:
Auditory stimuli have potential beneficial effects on cognitive functions and consciousness in patients with disorders of consciousness (DOC)，especially the emotional sound; however, precise and accurate quantitative indices to estimate cerebral activation to different auditory stimuli remain scarce. In this study, investigators assessed the response of different brain regions to three acoustic stimuli using quantitative electroencephalography (QEEG) and ERP(Event-related potential),and further investigated the predictive value of QEEG in the prognosis of DOC.

ELIGIBILITY:
Brain-damaged patients :

Inclusion Criteria:

1. Disorders of consciousness (Traumatic brain injury, stroke or anoxic encephalopathy)
2. Coma diagnosis (Plum and Posner, 1966), vegetative state (Task Force, 1994) or minimally conscious state (Giacino, Ashwal et al. 2002)
3. Lack of autonomic crisis since one week minimum
4. Medical condition considered stable
5. Patients who do not present hearing loss. Peaks I and II of Brainstem Auditory Evoked Potentials (BAEP) will be normal.

Exclusion Criteria:

1. hearing Problem
2. Uncontrolled Epilepsy
3. Autonomic crises
4. Medical unstable state
5. Pregnant or likely to be (interrogation data) or breastfeeding woman

Healthy participants :

Inclusion Criteria:

1. Subjects with normal hearing
2. Absence of neurological disorder
3. Subjects able to understand the experimental instructions

Exclusion Criteria:

1. Hearing problems and / or hearing loss higher than 30 decibels Hearing Level (dB HL) at a frequency band from 250 to 8000 Hz
2. Neurological disorders
3. Pregnant or likely to be (interrogation data) or breastfeeding woman

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
Glasgow Outcome Scale (GOS) | In one year
  A GOS value of <3 was considered as a bad recovery, while a GOS value of ≥3 was considered as a good recovery

SECONDARY OUTCOMES:
quantitative electroencephalography | 30 minutes before the auditory stimualtion and 30 minutes after each stimulation
  The power spectrum was divided into four bandwidths,an increase of delta and theta activity usually reflects encephalopathy and/or structural lesions, interpreted as poor outcome predictor of DOC. The power of α and β is related to the chance of recovery.

OTHER OUTCOMES:
N1,P300,LPP | From 200 msec before the stimuli onset to 1000ms after the auditory stimulation
  The event-related potential waveforms uncover voluntary responses to external stimuli that could assist in detecting signs of consciousness to reduce the risk of misdiagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Benyan Luo, Principal Investigator — The First Affiliated Hospital, Zhejiang University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu M, Bao WX, Zhang J, Hu YF, Gao J, Luo BY. Effect of acoustic stimuli in patients with disorders of consciousness: a quantitative electroencephalography study. Neural Regen Res. 2018 Nov;13(11):1900-1906. doi: 10.4103/1673-5374.238622. PMID 30233062